CLINICAL TRIAL: NCT01395004
Title: A Phase 2a, Open Label, Multicenter Study to Assess the Efficacy and Safety of the Oral AKT Inhibitor GSK2110183 in Subjects With Langerhans Cell Histiocytosis
Brief Title: A Study to Test the Ability of and Safety of GSK2110183 in Treating Langerhans Cell Histiocytosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 115397
Record Dates: First submitted 2011-07-12; First posted 2011-07-15 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Langerhans Cell Histiocytosis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — GSK2110183

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Drug - GSK2110183 (Experimental): This was an open-label study of oral GSK211083 administered at the maximum tolerated dose of 125 mg once daily.
  Interventions: Drug: GSK2110183

INTERVENTIONS:
Drug: GSK2110183 — GSK2110183 was orally administered at 125 mg once daily.

SUMMARY:
The purpose of this study was to assess safety and efficacy at months 3 and 6 in patients with Langerhans Cell Histiocytosis given daily oral doses of GSK2110183.

DETAILED DESCRIPTION:
LCH115397 was a phase 2a, open label, multicenter study testing 125 mg (starting dose) daily oral GSK2110183 in adult and adolescent patients with Langerhans Cell Histiocytosis. The primary objectives of the study were efficacy (at 3 and 6 months) and safety. For the purpose of efficacy analysis, patients were stratified into two groups: treatment-naïve (Stratum 1) and refractory or reactivation disease (Stratum 2). Adolescent participation was limited to patients with refractory or reactivation disease (Stratum 2).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is provided. Adolescents will provide assent, with consent provided by parent or legal guardian.
2. Prior therapy restrictions:

   * Refractory/reactivation stratum: Age >= 12 years of age at the time of study enrollment and Tanner Stage >2. Subjects less than 18 years old must weigh at least 40 kg.
   * Treatment-naïve stratum (defined as either no prior treatment or intolerant of first-line treatment with cessation prior to first response evaluation): Age >= 18 years old
3. Histologically- or cytologically-confirmed diagnosis of Langerhans Cell Histiocytosis requiring systemic treatment:

   * SS-LCH with 'CNS-risk' or 'special site' lesions or 'risk organs' (Includes LCH brain lesions or pituitary infiltration provided that disease is evaluable for treatment response. Patients with isolated pulmonary disease should have recent onset (within 3 years) or demonstrate evidence of active disease on PET or other functional imaging. If isolated pulmonary disease without radiographic lesion, then pulmonary function testing must demonstrate vital capacity <80% predicted, FEV1 <80% predicted or DLCO, <70% predicted, and condition is evaluable for treatment response and could not be explained through a diagnosis of asthma.)
   * SS-LCH with multifocal bone or skin disease
   * MS-LCH with or without involvement of 'risk organs'
4. Archival tumor available for central confirmation of LCH and biomarker analysis or willingness to undergo biopsy.
5. If 18 years or older, performance status score of 0, 1, and 2 according to the Eastern Cooperative Oncology Group (ECOG) scale. If age >=12 and <18, performance status score of >50 according to the Karnofsky performance status (KPS) scale.
6. Able to swallow and retain oral medication.
7. Male subjects with a female partner of childbearing potential must have had a prior vasectomy or agree to use adequate contraception from the time of the first dose of study drug until three months after the last dose of study drug.
8. A female subject is eligible to participate if she is of:

   * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/mL and estradiol < 40 pg/mL (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods defined in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least two to four weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
   * Child-bearing potential, has a negative serum pregnancy test during the screening period, and agrees to use adequate contraception from screening until four weeks after the last dose of study drug.

   Note: Oral contraceptives are not reliable due to potential drug-drug interaction.
9. Adequate organ-systems function.

Exclusion Criteria:

1. Chemotherapy, radiotherapy, or immunotherapy within 28 days (or 42 days for prior nitrosoureas or mitomycin C) prior to the first dose of study drug. Corticosteroids may be administered up to seven days prior to the first dose of study drug. Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity (in the medical opinion of the investigator) are permitted, if administered at least 14 days prior to the first dose of study drug.
2. Use of an investigational anti-cancer drug within 28 days or five half-lives, whichever is longer, preceding the first dose of GSK2110183.
3. Current use of a prohibited medication or requires any of these medications during treatment with GSK2110183.
4. Presence of active gastrointestinal disease or other condition that could affect gastrointestinal absorption (e.g. malabsorption syndrome) or predispose subject to gastrointestinal ulceration.
5. Any major surgery within the last four weeks (excluding diagnostic biopsy).
6. Unresolved toxicity (except alopecia) >= Grade 2 from previous therapy, except where the Investigator considers that the ongoing toxicity will not introduce additional risk factors and will not interfere with the study procedures.
7. Fasting serum glucose >126 mg/dL (7 mmol/L), or for known diabetic patients with stable disease, fasting serum glucose >250 mg/dL (14 mmol/L) and Hemoglobin A1c > 9%.
8. Current use of oral corticosteroids, with the exception of stress dose hydrocortisone (20 mg BID). Inhaled steroids permitted if patient is currently on a stable dose/regimen. Topical steroids are permitted; however, they should not be used as concurrent treatment for LCH skin disease.
9. Any serious or unstable pre-existing medical, psychiatric, or other condition (including lab abnormalities) that could interfere with subject safety or with obtaining informed consent.
10. Evidence of LCH-related neurodegenerative disease if patient has CNS SS-LCH, however, subjects with CNS SS-LCH who were previously treated for CNS involvement, and are currently asymptomatic without anti-epileptic medications or steroids for at least two months are eligible.
11. Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease).
12. Known infection with HIV, HBV or HCV.
13. QTc interval >= 470 msecs.
14. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within the past six months.
15. Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
16. Pregnant or lactating female.
17. History of previous treatment with a small molecule AKT inhibitor (this does not include perifosine), PI3K inhibitors, or mTOR inhibitors.
18. Other associated conditions which in the opinion of the investigator could significantly impair the ability to evaluate the impact of treatment on the clinical course of the disease.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Objective disease response at 3 and 6 months | Up to 6 months
Proportion of subjects experiencing greater than or equal to grade 3 neutropenia | Up to week 53
Proportion of patients who experience microbial infections | Up to week 53
Proportion of subjects experiencing newly diagnosed or worsening neuropathy | Up to week 53

CONTACTS AND LOCATIONS:
Overall Officials: Shannon R Morris, MD, PhD, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- See also: Results for study 115397 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115397?search=study&study_ids=115397#rs